CLINICAL TRIAL: NCT00428363
Title: Effect of Optic Edge Design in a Silicone Intraocular Lens on Posterior Capsule Opacification
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EK2512001
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2007-01-30 (Estimated); Status verified 2007-01

CONDITIONS: Cataract; Pseudophakia
Keywords: posterior capsule opacification; PCO; after cataract; intraocular lens; optic edge design; sharp optic edge
MeSH Terms: conditions — Cataract; Pseudophakia; Capsule Opacification | interventions — Cataract Extraction

INTERVENTIONS:
Device: Cataract surgery with implantation of an intraocular lens

SUMMARY:
Purpose: To compare the posterior capsule opacification (PCO) inhibiting effect of the sharp posterior optic edge design of the Clariflex silicone intraocular lens (IOL) with that of the double-round edge design of the SI40 (Phacoflex) silicone IOL over a period of 3 years.

Setting: Department of Ophthalmology, Medical University of Vienna, Vienna, Austria.

Methods: Fifty-two patients with bilateral age-related cataract (104 eyes) were included in this randomized, prospective, bilateral, patient- and examiner-masked clinical trial with intra-individual comparison. Each study patient had cataract surgery in both eyes and received an SI40 IOL (anterior and posterior round optic edges) in one eye and a Clariflex IOL with OptiEdge (round anterior and sharp posterior optic edge) in the other eye. Follow-up examinations were at one week, one month, six months, one, two, and three years. Digital retroillumination images were taken of each eye. The amount of PCO was assessed subjectively at the slit-lamp and objectively using automated image analysis software (AQUA) one, two, and three years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* bilateral, age related cataract

Exclusion Criteria:

* history of other ocular disease or intraocular surgery
* diabetes requiring medical control

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52
Dates: Start 2001-06; Study Completion 2006-03

PRIMARY OUTCOMES:
amount of posterior capsule opacification (objective and subjective score 0-10)

SECONDARY OUTCOMES:
visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Menapace, MD, Principal Investigator — Medical University of Vienna; Oliver Findl, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Dept. of Ophthalmology, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Buehl W, Findl O, Menapace R, Rainer G, Sacu S, Kiss B, Petternel V, Georgopoulos M. Effect of an acrylic intraocular lens with a sharp posterior optic edge on posterior capsule opacification. J Cataract Refract Surg. 2002 Jul;28(7):1105-11. doi: 10.1016/s0886-3350(02)01371-8. PMID 12106717
- [Background] Buehl W, Findl O, Menapace R, Sacu S, Kriechbaum K, Koeppl C, Wirtitsch M. Long-term effect of optic edge design in an acrylic intraocular lens on posterior capsule opacification. J Cataract Refract Surg. 2005 May;31(5):954-61. doi: 10.1016/j.jcrs.2004.09.053. PMID 15975461
- [Result] Buehl W, Menapace R, Sacu S, Kriechbaum K, Koeppl C, Wirtitsch M, Georgopoulos M, Findl O. Effect of a silicone intraocular lens with a sharp posterior optic edge on posterior capsule opacification. J Cataract Refract Surg. 2004 Aug;30(8):1661-7. doi: 10.1016/j.jcrs.2004.02.051. PMID 15313288